CLINICAL TRIAL: NCT01178047
Title: A Multicenter, Randomized, Double-blind Placebo Controlled Study to Assess the Effect of Rasagiline on Sleep-wake Disturbances in Patients With Parkinson's Disease (PD)
Brief Title: Multicenter Placebo Controlled Study to Assess the Effect of Rasagiline on Sleep-wake Disturbances in Patients With Parkinson's Disease
Acronym: Ras-PDS-1
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: payments stopped by grant provider
Sponsor: University of Zurich (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ras-PDS-1
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rasagiline (Active Comparator)
  Interventions: Drug: Rasagiline
- Placebo (Placebo Comparator)
  Interventions: Drug: Rasagiline

INTERVENTIONS:
Drug: Rasagiline — Rasagiline: 1 mg/d p.o. or Placebo one tablet p.o. once daily

SUMMARY:
Sleep-wake disturbances (SWD) are frequent in Parkinson's disease (PD) and affect the quality of life of affected patients.

Rasagiline is a potent, highly selective, irreversible, second-generation, monoamine oxidase type-B (MAO-B) inhibitor with a 24h dopaminergic effect.

It is well known that dopaminergic treatment closely interacts with SWD. This study aims to assess the effect of Rasagiline on SWD in PD patients. In this randomized, double-blind, placebo controlled study in clinical phase IV, 60 subjects will be treated with rasagiline 1mg po once daily or placebo over 8 weeks. The study is planned to be conducted in 6-9 Swiss centers. Questionaires will be used to assess SWDs: sleep disturbances (Parkinson's Disease Sleep Scale, PDSS), daytime sleepiness (Epworth Sleepiness Scale, ESS), fatigue (Fatigue Severity Scale, FSS), apathy (Apathy Evaluation Scale Self, AES-S), disability (Sheehan scale) and QoL in PD patients.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

1. Probable diagnosis of Parkinson's disease according to the modified UK Parkinson's Disease Society Brain Bank criteria
2. Hoehn and Yahr up to stage 3 in the off-state
3. Age = 40 years
4. On the basis of a physical examination and medical history, the patient is in the investigator's opinion otherwise healthy
5. Parkinson's Disease Sleep Scale (PDSS) score = 90.
6. Patients with stable dosage of hypnotics / sedative /neuropsychiatric treatment including antiParkinsonian treatment in the last 4 weeks before screening evaluation and with no change foreseen during the study period. Dose adjustments can be made, but no change or discontinuation of drugs.
7. Subjects must understand questionnaires in German, French or Italian
8. Provided signed informed consent
9. Females of childbearing potential must agree to utilize highly effective contraceptive methods of birth control.
10. Females of child bearing potential must have a negative pregnancy test.

Exclusion criteria:

1. Diagnosis unclear or suspicion of another than Parkinson's disease
2. Patients with cognitive deficit (MMSE < 26)
3. Patients who have undergone surgery for the treatment of PD
4. Patients with non-response to adequate antiParkinsonian treatment
5. History of moderate to severe hepatic insufficiency.
6. Clinically relevant or unstable vascular disease
7. History of drug or alcohol abuse (within the past 10 years)
8. Patients with a history of psychotic disorders
9. Patients with treatment resistant/recurrent major depression (HADS =19)
10. Patients with unstable dosage of antiParkinsonian or neuropsychiatric treatment in the last 4 weeks before screening evaluation.
11. Concomitant use of fluoxetine, fluvoxamine, pethidine or monoamine oxidase inhibitors (MAOI) during the course of the study and within 3 months prior to screening evaluation. Patient may be rescreened 3 months after discontinuation of the above mentioned drugs.
12. Concomitant use of dextromethorphan, ephedrine or pseudoephedrine during the course of the study
13. Women who are pregnant or lactating
14. Participation in another study during or up to 30 days prior to participation in this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of rasagiline on sleep disturbances in PD patients: Parkinson's Disease Sleep Scale (PDSS) | Baseline after 8 weeks of treatment
  Efficacy of rasagiline on sleep disturbances in PD patients: Parkinson's Disease Sleep Scale (PDSS)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Baumann, Assoc Prof, MD, Principal Investigator — University Hospital Zurich, Neurology
Locations (2):
- Switzerland (2):
  - University Hospital, Neurology, Zurich, Canton of Zurich
  - Neurocentro, Lugano, Lugano, Lugano